CLINICAL TRIAL: NCT03705806
Title: Evaluation of Toxicities With Thoracic Radiotherapy and Immune Checkpoint Inhibition in Non-small Cell Lung Cancer
Brief Title: Palliative Thoracic ImmunoRT
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 18-5327
Record Dates: First submitted 2018-08-15; First posted 2018-10-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer, Nonsmall Cell; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Study procedures include blood draw at baseline, end of radiation treatment, and at 1 month follow up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiation combined with immunotherapy — The trial is designed as a prospective observational single arm study investigating stage IV non-small cell lung cancer patients who are routinely treated with a PD-1 inhibitor for indications approved by Health Canada. All patients who are selected will be referred for palliative thoracic radiotherapy and treated with a standard dose prescription of 30 Gy in 10 fractions.

SUMMARY:
The trial is designed as a prospective observational single arm study investigating stage IV non-small cell lung cancer patients who are routinely treated with a PD-1 inhibitor for indications approved by Health Canada. All patients who are selected will be referred for palliative thoracic radiotherapy and treated with a standard dose prescription of 30 Gy in 10 fractions.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed AJCC 7th/8th edition Stage IV adenocarcinoma or squamous cell carcinoma not eligible for curative treatment.
2. Indication and suitability to receive palliative radiotherapy to the thorax (30Gy/10).
3. Receiving or planned to receive nivolumab or pembrolizumab
4. Prior history of systemic chemotherapy is permitted given a washout period of 4 weeks
5. Age 18 or older
6. ECOG Performance Status 0-2
7. Life expectancy greater than 3 months
8. Able and willing to provide informed consent
9. Able to complete patient reported outcome questionnaires

Exclusion Criteria:

1. Contraindications to radiotherapy, including a history of SLE, systemic scleroderma, IPF, ataxia telangiectasia
2. Previous history of thoracic radiotherapy with an overlapping field
3. Previous history of checkpoint inhibitor related pneumonitis or esophagitis
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include a population of patients with metastatic NSCLC on first or second line immunotherapy who have an indication for palliative thoracic radiation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Radiation related toxicities | up to 24 months
  rates of radiation-related toxicities in the combination of immunotherapy and palliative thoracic radiotherapy using CTCAE v5.0 grading
Patient Report Outcome | up to 12 months
  FACT-E
Patient experience and anxiety related to Quality of Life | up to 12 months
  EQ-5D

SECONDARY OUTCOMES:
Rate of Survival | 1 year
Rate of Survival | 2 year
Rate of Disease Recurrence | 3, 6, 12 months
  Patients will be followed for up to two years following the completion of their radiotherapy. They will undergo CT surveillance imaging as standard by routine immunotherapy protocol with a minimum of 3 scans at the 3, 6 and 12 month mark. Local and distant recurrence will be determined primarily by CTCAE with CT scans as per ir-RECIST v1.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No